CLINICAL TRIAL: NCT06377280
Title: An Un-controlled, Prospective, Multi-center, Post Market Clinical Follow-up Investigation to Confirm Performance and Safety of Navina Mini, a New CE-marked Low-volume Transanal Irrigation (TAI) Device.
Brief Title: En Evaluation of Navina Mini, a New Low-volume Transanal Irrigation Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAV-0011
Record Dates: First submitted 2023-09-28; First posted 2024-04-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): The investigational subjects are persons with anal incontinence or outlet problems and deemed suitable for and in need of low-volume TAI as assessed by the investigator or designee
  Interventions: Device: Navina Mini

INTERVENTIONS:
Device: Navina Mini — CE-marked Navina Mini, released on the market May 2023

SUMMARY:
This is an un-controlled, prospective, multi center, post market clinical follow-up investigation that will enroll male and female subjects in need of bowel management with low-volume transanal irrigation (TAI) as judged by the investigator. A total of 40 investigational subjects in need of low-volume TAI will be recruited from 2-3 sites in Sweden and will be treated with Navina Mini as per product intended purpose and per instruction of use during a period of four weeks.

Participating subjects will perform three visits during the clinical investigation and will be followed for a total of four weeks. The first visit, Visit 1, will be performed at the investigational clinic to assess eligibility, collect demographics, baseline data and instruct how to use the device. Visit 2 will be performed after two weeks of treatment through telephone contact. The final visit, Visit 3, will be performed after additional two weeks of treatment, and can be performed either at the investigational clinic or through telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Anal incontinence or faecal outlet problems without any pathological obstruction in the ano-rectum.
* Symptom duration of > 6 months
* Adult male and females >18 years old
* Patient can communicate in written and oral Swedish language

Exclusion Criteria:

* Subjects treated with high volume TAI i.e., volume > 250 ml
* Pregnancy at the time of enrollment
* Participating in another clinical investigation interfering with this investigation
* Subjects with active, symptomatic inflammatory bowel disease, radiation proctitis and or active perianal fistula disease
* Rectal bleeding of uncertain origin or active hemorrhoidal bleeding
* < 6 months after anal or colorectal surgery
* Ongoing anti-coagulant therapy (eg. NOACS, heparin, Warfarin)
* Acute diverticulitis and diverticular abscess
* Ischemic colitis
* Colorectal cancer
* Any physical handicap that prevents usage of product
* Inability to use product or anyone to assist in its usage
* Person not suitable for the investigation according to the investigator judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 4 weeks
  Patient Reported Outcome - Overall patient satisfaction when performing low- volume trans-anal irrigation measured with a 5-graded scale [0 = Not at all satisfied, 1 = Not satisfied, 2 = Neither satisfied nor unsatisfied, 3=Satisfied, 4 = Very satisfied]

SECONDARY OUTCOMES:
Assessment of clinical benefit | 4 weeks
  Patient Reported Outcome on Fecal Incontinence and Defecation syndrome
Ease of handling | 4 weeks
  Patient Reported Outcome on perception of handling the device
Safety Outcome | 4 weeks
  Assessment of adverse events and device deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Louis Banka Johnson, MD, Principal Investigator — University Hospital of Malmö, Sweden
Locations (1):
- Skåne University Hospital, Malmo, Sweden